CLINICAL TRIAL: NCT02750189
Title: The Economic Burden of Patients With COPD in South Korea
Brief Title: The Economic Burden of Chronic Obstructive Pulmonary Disease(COPD) in South Korea
Acronym: BOC
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kwang-Ha Yoo, Professor, Konkuk University Medical Center
Other Study IDs: KUH1010636
Record Dates: First submitted 2016-03-28; First posted 2016-04-25 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Direct Service Costs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Mild Group: FEV₁/FVC <70% and FEV₁≥80% direct/indirect cost
  Interventions: Other: Direct cost; Other: Indirect cost
- Moderate Group: FEV₁/FVC <70% and 50%≤FEV₁≤80% direct/indirect cost
  Interventions: Other: Direct cost; Other: Indirect cost
- Severe Group: FEV₁/FVC <70% and 30%≤FEV₁≤50% direct/indirect cost
  Interventions: Other: Direct cost; Other: Indirect cost
- Very Severe Group: FEV₁/FVC <70% and FEV₁<30% direct/indirect cost
  Interventions: Other: Direct cost; Other: Indirect cost

INTERVENTIONS:
Other: Direct cost — Money spent to treat COPD in medical institute based on HIRA
Other: Indirect cost — extra-expanses excluding hospital fees

SUMMARY:
The purpose of this study is to estimate a direct/indirect medical cost and to provide evidence establishing efficient strategies to reduce medical costs of COPD in Korea.

DETAILED DESCRIPTION:
This study is a multi-center research on economic burdens of COPD for a year. It is composed of three phases detailed as follow.

Phase 1: Direct Cost Estimation in COPD patients (N = 400) Direct cost determined as amount of money expended to medical institutes for treatment. Estimated costs, based on the information from Health insurance review agency(HIRA) and The National Health and Nutrition Examination Survey (NHANES) data, are collected.

Phase 2: Indirect cost Estimation by Sampling Survey in COPD patient Indirect cost is extra-expanses excluding hospital fees, including cost for transportation, medical instruments, home care services and loss of labor capacity reduction. The information was collected by structured questionnaire for 12 weeks.

Phase 3: Direct/Indirect cost is validated and analyzed based on the collected information from phase 1 and 2 according to severity defined by the GOLD guideline.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* COPD patients

Exclusion Criteria:

* Patients who disagree with participating in research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease (COPD)
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Total cost of COPD | 1 year
  Korean won, KRW

SECONDARY OUTCOMES:
The number of acute exacerbations | 1 year
  Number of events
The cost of alternative medication use | three months
  We will add up the costs of herbal medicine, health supplement, medical equipments and respiratory rehabilitation. According to patients, the items of alternative medication use would be different.
Cost of productivity lost | Last 7days from filling out questionnaires
  Reduction of working hour and monthly income for being late or abscence from work.
EuroQol five dimension(EQ-5D) | 3 months
  Measured by questionnaire based by EQ -5D ( EQ-5D essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) . The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems )
The total number of visits | 1 year
  primary clinics, emergency department and hospital admission.
Nursing cost | 1 year (past 1 year before filling questionnaires)
  payment for nurse (Korean won, KRW)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Ha NA Yoo, Doctor, Principal Investigator — Konkuk University Hospial
Locations (1):
- Konkuk University Hospital, Gwangjin Gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guarascio AJ, Ray SM, Finch CK, Self TH. The clinical and economic burden of chronic obstructive pulmonary disease in the USA. Clinicoecon Outcomes Res. 2013 Jun 17;5:235-45. doi: 10.2147/CEOR.S34321. Print 2013. PMID 23818799
- [Background] Dang-Tan T, Ismaila A, Zhang S, Zarotsky V, Bernauer M. Clinical, humanistic, and economic burden of chronic obstructive pulmonary disease (COPD) in Canada: a systematic review. BMC Res Notes. 2015 Sep 21;8:464. doi: 10.1186/s13104-015-1427-y. PMID 26391471
- [Background] Lokke A, Hilberg O, Tonnesen P, Ibsen R, Kjellberg J, Jennum P. Direct and indirect economic and health consequences of COPD in Denmark: a national register-based study: 1998-2010. BMJ Open. 2014 Jan 6;4(1):e004069. doi: 10.1136/bmjopen-2013-004069. PMID 24394800
- [Background] Sullivan SD, Ramsey SD, Lee TA. The economic burden of COPD. Chest. 2000 Feb;117(2 Suppl):5S-9S. doi: 10.1378/chest.117.2_suppl.5s. PMID 10673466
- [Background] Mannino DM, Higuchi K, Yu TC, Zhou H, Li Y, Tian H, Suh K. Economic Burden of COPD in the Presence of Comorbidities. Chest. 2015 Jul;148(1):138-150. doi: 10.1378/chest.14-2434. PMID 25675282
- [Background] Teo WS, Tan WS, Chong WF, Abisheganaden J, Lew YJ, Lim TK, Heng BH. Economic burden of chronic obstructive pulmonary disease. Respirology. 2012 Jan;17(1):120-6. doi: 10.1111/j.1440-1843.2011.02073.x. PMID 21954985
- [Background] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Background] Kim J, Lee TJ, Kim S, Lee E. The economic burden of chronic obstructive pulmonary disease from 2004 to 2013. J Med Econ. 2016;19(2):103-10. doi: 10.3111/13696998.2015.1100114. Epub 2015 Oct 19. PMID 26414920
- See also: Health insurance review agency in south korea — http://www.hira.or.kr/main.do